CLINICAL TRIAL: NCT04141774
Title: Stroke Rehabilitation Using BCI Technology
Brief Title: Stroke Rehabilitation Using Brain-Computer Interface (BCI) Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0971; 1R01NS105646-01A1 (NIH); A539300 (Other: UW Madison); SMPH/RADIOLOGY (Other: UW Madison); Protocol Version 2/1/22 (Other: UW Madison)
Record Dates: First submitted 2019-10-15; First posted 2019-10-28 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: aneurysm; transient ischemic attack
MeSH Terms: conditions — Stroke; Aneurysm; Ischemic Attack, Transient | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Passive FES (Active Comparator): Subjects randomized to this control group will be asked to participate in a passive FES intervention or non-EEG guided muscle stimulation. Participation will include behavioral assessments, functional magnetic resonance imaging, and functional electric stimulation (FES) treatment.
  Interventions: Device: Functional Electric Stimulation (FES); Behavioral: Behavioral Assessments; Other: Magnetic Resonance Imaging
- Active FES (Experimental): Subjects randomized to this experimental group will be asked to complete the active FES intervention which include EEG guided muscle stimulation. Participation will include behavioral assessments, functional magnetic resonance imaging, functional electric stimulation (FES) treatment, and EEG.
  Interventions: Device: Functional Electric Stimulation (FES); Behavioral: Behavioral Assessments; Other: Magnetic Resonance Imaging; Other: EEG

INTERVENTIONS:
Device: Functional Electric Stimulation (FES) — FES uses low energy electrical pulses to artificially generate body movements in individuals with muscle paralysis. FES can be used to generate muscle contraction in otherwise paralyzed limbs to restore function.
Behavioral: Behavioral Assessments — These assessments will include measures of upper extremity motor assessments, standard stroke scales, and measures of activities of daily living.
Other: Magnetic Resonance Imaging — A functional magnetic resonance image will be collected.
Other: EEG — EEG electrodes will be attached to the subject's scalp using a standard, commercially available electrode cap. Proper electrode placement is made according to the international 10-20 system, ensuring complete electrode coverage over sensorimotor cortex.
  Other Names: Electroencephalography
  Arms: Active FES

SUMMARY:
The purpose of this research is to determine if functional muscle stimulation, directed by electroencephalogram (EEG) output, can increase the extent of stroke recovery on behavioral measures and induce brain plasticity as measured by functional magnetic resonance imaging (fMRI). Participants will include stroke patients with upper-limb hemiparesis and can expect to be on study for approximately 4 months.

DETAILED DESCRIPTION:
Ongoing research (NCT02098265) suggests that noninvasive EEG driven Brain Computer Interface (BCI) systems hold the potential for facilitating recovery in the chronic phase after stroke by synchronizing central or brain activity with peripheral movements and thereby harnessing brain plasticity.

The specific aims of this study are:

Aim 1: To investigate the efficacy of active FES vs. passive FES, as measured by changes in behavioral measures. The investigators hypothesize that improvements in motor function will be significantly greater using the active FES therapy than the passive FES therapy.

Aim 2: To investigate the relationship between brain functional activation patterns and behavior changes induced by active vs. passive FES intervention. The investigators hypothesize that changes induced by active FES (as measured by brain fMRI and EEG measures) will show greater adaptive brain reorganization changes (i.e. brain changes that correlate with improved outcomes) than that induced by the passive FES.

Aim 3: To investigate the relationship between brain white matter integrity and behavior changes induced by active vs. passive FES intervention. The investigators hypothesize that changes induced by active FES (as measured by brain DTI measures) will show greater adaptive brain reorganization changes (i.e. brain changes that correlate with improved outcomes) than that induced by the passive FES.

ELIGIBILITY:
Inclusion Criteria:

* New-onset ischemic stroke 12 months prior - chronic time frame;
* Right hand dominant - affected arm;
* Mild to moderate unilateral upper extremity impairment or severe unilateral upper extremity impairment;
* No upper extremity injury or conditions that limited use prior to the stroke;
* Must be able to provide informed consent on their own behalf.

Exclusion Criteria:

* Inability to competently participate in study procedures
* Concurrent upper extremity therapy, other neurological or psychiatric disorders

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Prabhakaran, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Young BM, Stamm JM, Song J, Remsik AB, Nair VA, Tyler ME, Edwards DF, Caldera K, Sattin JA, Williams JC, Prabhakaran V. Brain-Computer Interface Training after Stroke Affects Patterns of Brain-Behavior Relationships in Corticospinal Motor Fibers. Front Hum Neurosci. 2016 Sep 16;10:457. doi: 10.3389/fnhum.2016.00457. eCollection 2016. PMID 27695404
- [Result] Young BM, Nigogosyan Z, Walton LM, Remsik A, Song J, Nair VA, Tyler ME, Edwards DF, Caldera K, Sattin JA, Williams JC, Prabhakaran V. Dose-response relationships using brain-computer interface technology impact stroke rehabilitation. Front Hum Neurosci. 2015 Jun 23;9:361. doi: 10.3389/fnhum.2015.00361. eCollection 2015. PMID 26157378
- [Result] Song J, Nair VA, Young BM, Walton LM, Nigogosyan Z, Remsik A, Tyler ME, Farrar-Edwards D, Caldera KE, Sattin JA, Williams JC, Prabhakaran V. DTI measures track and predict motor function outcomes in stroke rehabilitation utilizing BCI technology. Front Hum Neurosci. 2015 Apr 27;9:195. doi: 10.3389/fnhum.2015.00195. eCollection 2015. PMID 25964753
- [Result] Song J, Young BM, Nigogosyan Z, Walton LM, Nair VA, Grogan SW, Tyler ME, Farrar-Edwards D, Caldera KE, Sattin JA, Williams JC, Prabhakaran V. Characterizing relationships of DTI, fMRI, and motor recovery in stroke rehabilitation utilizing brain-computer interface technology. Front Neuroeng. 2014 Jul 29;7:31. doi: 10.3389/fneng.2014.00031. eCollection 2014. PMID 25120466
- [Result] Young BM, Nigogosyan Z, Nair VA, Walton LM, Song J, Tyler ME, Edwards DF, Caldera K, Sattin JA, Williams JC, Prabhakaran V. Case report: post-stroke interventional BCI rehabilitation in an individual with preexisting sensorineural disability. Front Neuroeng. 2014 Jun 24;7:18. doi: 10.3389/fneng.2014.00018. eCollection 2014. PMID 25009491
- See also: Publication resulting from this work. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5025476/
- See also: Publication resulting from this work. — https://www.ncbi.nlm.nih.gov/pubmed/26157378
- See also: Publication resulting from this work. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4410488/
- See also: Publication resulting from this work. — https://www.ncbi.nlm.nih.gov/pubmed/25120466
- See also: Publication resulting from this work. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4067954/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Passive FES | Active FES
Started | 42 | 42
Baseline 1 (Pre-intervention) | 42 | 42
Baseline 2 (Pre-intervention, Approximately 1 Month From Baseline 1) | 42 | 42
7 Weeks (Mid-intervention) | 41 | 40
10 Weeks (End of Intervention) | 40 | 42
4 Months (Post-intervention) | 41 | 41
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Passive FES | Active FES | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Full Range); unit: years] | 67.38 [54 to 82] | 66.67 [53 to 80] | 67.03 [53 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 24 | 21 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 42 | 41 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 40 | 38 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Action Research Arm Test Scores
Description: The Action Research Arm Test (ARAT) is designed for evaluation of upper extremity function. This test consists of sections for Grasp, Grip, Pinch and Gross Movements and comprise a total of 19 tests. Each test is scored 0-3 where 0 is 'no movement' and 3 is 'the movement is performed normally'. Each section is scored separately and the scores added for a total possible range of scores from 0-57 where the higher the score, the complete and efficient the movement. Scores will be reported for baseline, mid (~7 weeks), post (~10 weeks), and end of study, up to 4 months.
Time Frame: baseline, 7 weeks, 10 weeks, 4 months
Population: Some participants did not provide data for all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 42 | 42
score on a scale
  baseline | 28.10 (17.84) | 27.76 (18.38)
  7 weeks: number analyzed (Participants) | 41 | 40
  7 weeks | 29.95 (17.30) | 30.18 (18.30)
  10 weeks: number analyzed (Participants) | 40 | 42
  10 weeks | 32.53 (16.97) | 32.83 (18.60)
  4 months: number analyzed (Participants) | 41 | 41
  4 months | 31.78 (16.85) | 34.10 (18.57)

2. Primary Outcome: Stroke Impact Scale
Description: The Stroke Impact Scale, or SIS, was created to assess changes in impairments, activities and participation following a stroke. Scores on the SIS will provide an index of clinically "meaningful" change representing the change in the patient's mental and physical abilities concurrent with their performance on the verbal fluency and memory tasks. The 4 physical function domains (strength, hand function, activities of daily living (ADL)/instrumental activities of daily living (IADL), and mobility) will be collapsed to a physical function subscale. All domain scores range from 0 to 100 with 100 being the best.
Time Frame: baseline, 7 weeks, 10 weeks, 4 months
Population: Some participants did not provide data at all timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 42 | 42
score on a scale
  baseline | 61.90 (24.68) | 66.07 (23.32)
  7 weeks: number analyzed (Participants) | 41 | 40
  7 weeks | 70.29 (19.81) | 68.22 (22.00)
  10 weeks: number analyzed (Participants) | 40 | 42
  10 weeks | 69.97 (22.64) | 67.35 (21.24)
  4 months: number analyzed (Participants) | 41 | 41
  4 months | 59.86 (14.50) | 78.49 (14.61)

3. Secondary Outcome: Change in Electroencephalogram (EEG) Response Strength
Description: EEG was recorded in microvolts (µV) from electrodes C4/C3 during periods of left arm imagery and right arm imagery. EEG Response strength is defined as the spectral power in the mu + beta frequency band (8-30 Hz), averaged over the BCI trials. For each participant and time point, a ratio was computed: Ratio = Power_Left Imagery / Power_Right Imagery.
Time Frame: baseline 1, baseline 2, 7 weeks, 10 weeks, 4 months
Population: Some participants did not provide data at all time points
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 42 | 42
ratio
  Baseline 1 | 1.120 (0.119) | 0.882 (0.090)
  Baseline 2 | 0.855 (0.228) | 1.145 (0.126)
  7 weeks: number analyzed (Participants) | 41 | 40
  7 weeks | 0.970 (0.205) | 1.236 (0.113)
  10 weeks: number analyzed (Participants) | 40 | 42
  10 weeks | 0.957 (0.171) | 1.328 (0.234)
  4 months: number analyzed (Participants) | 41 | 41
  4 months | 1.125 (0.131) | 1.228 (0.083)

4. Secondary Outcome: Signal Change in Functional Magnetic Resonance Imaging (MRI)
Description: To compare the percent signal change in the functional MRI activations before and after functional stimulation.
Time Frame: baseline 1, baseline 2, 7 weeks, 10 weeks, 4 months
Population: Some participants did not provide data at all time points
Measure: Mean (Standard Deviation); unit: percent signal change
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 42 | 42
percent signal change
  Baseline 1 | 1.136 (0.466) | 1.203 (0.461)
  Baseline 2 | 1.003 (0.459) | 1.153 (0.440)
  7 weeks: number analyzed (Participants) | 41 | 40
  7 weeks | 1.130 (0.518) | 1.108 (0.461)
  10 weeks: number analyzed (Participants) | 40 | 42
  10 weeks | 1.117 (0.581) | 1.156 (0.583)
  4 months: number analyzed (Participants) | 41 | 41
  4 months | 1.121 (0.423) | 1.192 (0.482)

5. Secondary Outcome: Nine Hole Peg Test (9HPT)
Description: The 9-HPT is a quick and easy to administer tool for screening fine motor problems in participants. It is a timed test in which nine pegs are inserted and removed from nine holes in the pegboard with each hand. Measured at 5 time points over the length of the study.
Time Frame: baseline 1, baseline 2, 7 weeks, 10 weeks, 4 months
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 42 | 42
seconds
  Baseline visit 1 | 59.89 (4.780) | 59.07 (4.656)
  Baseline visit 2 | 59.53 (4.629) | 59.24 (4.676)
  7 weeks: number analyzed (Participants) | 41 | 40
  7 weeks | 59.65 (3.681) | 58.52 (5.066)
  10 weeks: number analyzed (Participants) | 40 | 42
  10 weeks | 59.07 (5.047) | 58.64 (5.565)
  4 months: number analyzed (Participants) | 41 | 41
  4 months | 58.15 (5.236) | 56.29 (3.935)

6. Secondary Outcome: Motor Activity Log (MAL): Amount of Use
Description: The MAL is a structured interview developed to assess the use of the more affected upper extremity (UE) in real-world daily activities. Assessed at 5 time points over the length of the study. The Amount of Use scoring is as follows (intermediate scores are possible, 0.5 between each whole number):
  * 0 - Did not use my weaker arm (not used).
  * 1 - Occasionally used my weaker arm, but only very rarely (very rarely).
  * 2 - Sometimes used my weaker arm but did the activity most of the time with my stronger arm (rarely).
  * 3 - Used my weaker arm about half as much as before the stroke (half pre-stroke).
  * 4 - Used my weaker arm almost as much as before the stroke (3/4 pre-stroke).
  * 5 - Used my weaker arm as often as before the stroke (same as pre-stroke).
Time Frame: baseline 1, baseline 2, 7 weeks, 10 weeks, 4 months
Population: Some participants did not provide data at all timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 42 | 42
score on a scale
  baseline 1 | 0.9888 (0.3004) | 1.280 (0.3071)
  baseline 2 | 1.052 (0.2902) | 1.452 (0.3665)
  7 weeks: number analyzed (Participants) | 41 | 40
  7 weeks | 1.413 (0.3252) | 1.750 (0.2934)
  10 weeks: number analyzed (Participants) | 40 | 42
  10 weeks | 1.631 (0.2813) | 2.048 (0.2766)
  4 months: number analyzed (Participants) | 41 | 41
  4 months | 1.750 (0.3137) | 2.603 (0.3151)

7. Secondary Outcome: Motor Activity Log (MAL): Quality of Movement
Description: The MAL is a structured interview developed to assess the use of the more affected upper extremity (UE) in real-world daily activities. Assessed at 5 time points over the length of the study. The Quality of Movement was scored as follows (intermediate scores 0.5 between whole numbers are possible):
  * 0 - The weaker arm was not used at all for that activity (never).
  * 1 - The weaker arm was moved during that activity but was not helpful (very poor).
  * 2 - The weaker arm was of some use during that activity but needed some help from the stronger arm or moved very slowly or with difficulty (poor).
  * 3 - The weaker arm was used for the purpose indicated but movements were slow or were made with only some effort (fair).
  * 4 - The movements made by the weaker arm were almost normal, but were not quite as fast or accurate as normal (almost normal).
  * 5 - The ability to use the weaker arm for that activity was as good as before the stroke (normal).
Time Frame: baseline 1, baseline 2, 7 weeks, 10 weeks, 4 months
Population: Some participants did not provide data at all timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 42 | 42
score on a scale
  baseline 1 | 0.9564 (0.2786) | 1.219 (0.3305)
  baseline 2 | 1.073 (0.3130) | 1.372 (0.3690)
  7 weeks: number analyzed (Participants) | 41 | 40
  7 weeks | 1.363 (0.3600) | 1.846 (0.2713)
  10 weeks: number analyzed (Participants) | 40 | 42
  10 weeks | 1.557 (0.2645) | 2.164 (0.3438)
  4 months: number analyzed (Participants) | 41 | 41
  4 months | 1.854 (0.2726) | 2.541 (0.3480)

8. Secondary Outcome: Change in Modified Ashworth Scale (MAS)
Description: The MAS measures spasticity where 0 is no increase in muscle tone to 4 where affected part is in rigid in flexion or extension. Assessed at 5 time points over the length of the study.
Time Frame: 4 months
Population: MAS data were not collected in order to reduce participant burden associated with completing multiple assessments during study visits. The protocol was not amended to reflect this.
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Hand Grip Strength
Description: Hand Grip Strength will be assessed using a dynamometer. Measured at 5 time points over the length of the study.
Time Frame: baseline 1, baseline 2, 7 weeks, 10 weeks, 4 months
Population: Some participants did not provide data at all timepoints.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 42 | 42
kilograms
  baseline 1 | 32.95 (18.69) | 31.54 (18.61)
  baseline 2 | 32.86 (19.01) | 31.10 (18.82)
  7 weeks: number analyzed (Participants) | 41 | 40
  7 weeks | 34.66 (18.11) | 34.78 (17.92)
  10 weeks: number analyzed (Participants) | 40 | 42
  10 weeks | 37.45 (17.43) | 37.29 (18.56)
  4 months: number analyzed (Participants) | 41 | 41
  4 months | 37.37 (16.68) | 38.68 (17.32)

10. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)
Description: The CES-D is a self-report scale and includes 20 items that survey mood, somatic complaints, interactions with others, and motor functioning in the past week. Total possible score 0-60, with the higher score indicating more symptoms of depression. Assessed at 5 time points over the length of the study.
Time Frame: 4 months
Population: CES-D data were not collected in order to reduce participant burden associated with completing multiple assessments during study visits. The protocol was not amended to reflect this.
Arm/Group | Passive FES | Active FES
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 4 months
Arm/Group | Passive FES | Active FES
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04141774/Prot_SAP_000.pdf